CLINICAL TRIAL: NCT01891032
Title: Assessment of Acute Renal Injury During Partial Nephrectomy Using Neutrophil Gelatinase-associated Lipocalin (NGAL): Prospective Comparative Study Between Open, Video-assisted Minilaparotomy, Laparoscopic, and Robotic-assisted Laparoscopic Surgery
Status: Completed | Type: Observational
Sponsor: Yonsei University (Other)
Responsible Party: Sponsor
Other Study IDs: 4-2013-0261
Record Dates: First submitted 2013-06-27; First posted 2013-07-02 (Estimated); Last update posted 2014-07-28 (Estimated); Status verified 2014-07

CONDITIONS: the Patients With Partial Nephrectomy
Keywords: acute kidney injury, partial nephrectomy, biomarker
MeSH Terms: conditions — Acute Kidney Injury

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (4):
- the patients with open partial nephrectomy: the adult patients with open partial nephrectomy
- laparoscopic: the adult patients with laparoscopic partial nephrectomy
- VAMS: the adult patients with VAMS partial nephrectomy
- robotic: the adult patients with robotic partial nephrectomy

SUMMARY:
Urinary Neutrophil gelatinase associated lipocalin (NGAL) has been recently reported to be related with the degree of acute kidney injury. We are trying to analyze whether it is related with the grade of acute kiney injury after partial nephrectomy and there is any difference between the kinds of surgery.

ELIGIBILITY:
Inclusion Criteria:

1. adults patient more than 20 years old with ASA score 1-3
2. the patients who undergoing partial nephrectomy for the renal mass less than 7 cm

Exclusion Criteria:

1. the patient with previous history with renal surgery
2. the patient with bilateral partial nephrectomy
3. the patient with synchronous operation for other intraperitoneal surgery
4. the renal mass more than 7 cm
5. previous kinds of surgery is changed into other kinds due to bleeding, etc
6. the patient with serum Cr level more than 1.4 mg/dl
7. the patient who does not understand the consent form

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 1. the adult patients with open partial nephrectomy
  2. the adult patients with laparoscopic partial nephrectomy
  3. the adult patients with VAMS partial nephrectomy, 4: the adult patients with robotic partial nephrectomy
Sampling Method: Non-Probability Sample
Enrollment: 160 (Actual)
Dates: Start 2013-06; Primary Completion 2014-04 (Actual); Study Completion 2014-05 (Actual)

PRIMARY OUTCOMES:
The level of urinary NGAL | changes from Preoperative, postop 3hr, 24hr, 48hrs after partial nephrectomy
  Analysis of correlation between the level of preoperative and postoperative urinary NGAL

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Urology, Urological Science Institute, Yonsei University, Colleage of Medicine, Seoul, Seoul, South Korea